CLINICAL TRIAL: NCT00475956
Title: Phase I, Open-Label Study To Assess the Safety, Tolerability and Pharmacokinetics of Daily Oral Doses of Cediranib (RECENTIN™;AZD2171) (20, 30 or 45mg) When Co-Administered With Daily Oral Doses of AZD0530 (125mg or 175mg) in Patients With Advanced Solid Tumours
Brief Title: Safety and Tolerability Study of AZD2171 in Combination With AZD0530 in Patients With Advanced Solid Tumours
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Jane Robertson, MSD, AstraZeneca
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D8480C00014; EuDract #2006-003505-55
Record Dates: First submitted 2007-05-18; First posted 2007-05-21 (Estimated); Last update posted 2010-04-15 (Estimated); Status verified 2010-04

CONDITIONS: Neoplasms
Keywords: Cancer; Tumour; Advanced Solid Tumour; Lung Cancer; Breast Cancer; Cholangiocarcinoma; Colon Cancer; Gastric Cancer; Choriocarcinoma; Liver Cancer; Myeloma; Ovarian Cancer; Pancreatic Cancer; Peritoneal Cancer
MeSH Terms: conditions — Neoplasms; Lung Neoplasms; Breast Neoplasms; Cholangiocarcinoma; Colonic Neoplasms; Stomach Neoplasms; Choriocarcinoma; Liver Neoplasms; Neoplasms, Plasma Cell; Ovarian Neoplasms; Pancreatic Neoplasms | interventions — cediranib; saracatinib

ARMS (2):
- 1 (Experimental): AZD2171 Monotherapy
  Interventions: Drug: AZD2171
- 2 (Experimental): AZD2171 + AZD0530
  Interventions: Drug: AZD2171; Drug: AZD0530

INTERVENTIONS:
Drug: AZD2171 — oral tablet multiple ascending doses 20, 30 or 45 mg
  Other Names: cediranib; RECENTIN™
Drug: AZD0530 — oral tablet multiple ascending doses 125 mg or 175 mg
  Arms: 2

SUMMARY:
The purpose of the study is to determine if the maximum tolerated doses of AZD2171, in combination with AZD0530, in treating patients with advanced solid tumours are safe, tolerable and efficacious.

ELIGIBILITY:
Inclusion Criteria:

* Written consent
* Cancer diagnosis & stage
* Patients for whom no standard therapy exists
* World Health Organization (WHO) performance status 0-2
* One or more measurable lesions

Exclusion Criteria:

* Prostate cancer
* Untreated unstable brain or meningeal metastases
* Specific laboratory ranges
* Pregnant or breast-feeding women
* Any evidence of severe or uncontrolled diseases
* Participation in other trials within 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-05; Primary Completion 2008-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Determine the safety and tolerability of ascending daily oral doses of AZD2171 when co-administered with AZD0530 to patients with advanced solid tumours by assessment of AEs, vital signs, HRCT Scans, clin chem, haematology, urinalysis, ECG and phys exam | assessed at each visit

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of AZD2171 alone and in combination with AZD0530 | assessed at each visit
Safety and efficacy | assessed at each visit
Genetic variation of pathways targeted by AZD2171 and AZD0530 | assessed during study

CONTACTS AND LOCATIONS:
Overall Officials: Jane Roberston, Study Director — AstraZeneca; Tanja Trarbach, MD, Principal Investigator — Universitatsklinikum der GHS Essen
Locations (3):
- Germany (3):
  - Research Site, Freiburg im Breisgau, Baden-Wurttemberg
  - Research Site, Essen, Ruhr
  - Research Site, Herne, Ruhr